CLINICAL TRIAL: NCT01597830
Title: The Effects of Specialized Footwear in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Najia Shakoor, M.D., Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L07041071
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; loading
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active shoe (Experimental)
  Interventions: Other: Mobility shoe
- Control (Sham Comparator)
  Interventions: Other: control shoe

INTERVENTIONS:
Other: Mobility shoe — flat, specialized shoe
  Arms: active shoe
Other: control shoe — control shoe
  Arms: Control

SUMMARY:
This study evaluates the effects of specialized footwear on pain and knee loading in knee osteoarthritis. The hypothesis is that this footwear will lead to decreased knee loading and knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent and to comply with the study protocol and follow-up instructions.
* Symptomatic OA of the knee, as defined by the American College of Rheumatology's Clinical Criteria for Classification and Reporting of OA of the Knee. If symptoms are bilateral, then the knee identified by the subject as more symptomatic will serve as the index knee.
* Ambulatory knee pain, defined as the presence of greater than 30 mm of pain while walking on a flat surface (corresponding to question 1 of the visual analog format of the WOMAC.
* Radiographic OA of the study knee of grade 2 or 3, as defined by the modified Kellgren and Lawrence (K-L) grading scale.
* Medial compartment OA, defined as either qualitative joint space narrowing of ≥ 1or the presence of medial bone cyst, sclerosis, or osteophyte.

Exclusion Criteria:

* Inability or unwillingness to wear study shoes for at least 6 hours/day for 6 days/week
* Knee flexion contracture of > 15 degrees or inability to ambulate without assistance.
* Presence of clinically significant OA of the hip or ankle or pain greater than 20 mm at these sites (WOMAC).
* > 3 degrees valgus or >12 degrees varus deformity of either knee, defined by the mechanical axis (hip-knee angle).
* Predominant lateral compartment OA, defined as narrowing of the lateral joint space in excess of the narrowing of the medial joint space in either the index or the contralateral knee.
* Concurrent systemic inflammatory arthropathy,
* Prior knee or hip arthroplasty, or surgical arthroscopy of either knee within previous 3 months or history of fracture of either lower extremity within 6 months of study entry.
* Intrinsic foot disease including hallux rigidus, hallux abducto-valgus, metatarsalgia, plantar fasciitis, peripheral neuropathy, or any foot condition that may be exacerbated by particular footwear.
* Intra-articular injection in the index knee: steroids within 6 weeks, hyaluronan derivatives within 4 months.
* Pregnant subjects will be excluded because of the X-rays required.
* Any medical condition that, in the opinion of the PI, would render the subject unable to complete the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-07; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Dynamic knee loading | 6 months to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Najia Shakoor, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Shakoor N, Sengupta M, Foucher KC, Wimmer MA, Fogg LF, Block JA. Effects of common footwear on joint loading in osteoarthritis of the knee. Arthritis Care Res (Hoboken). 2010 Jul;62(7):917-23. doi: 10.1002/acr.20165. PMID 20191571
- [Background] Shakoor N, Lidtke RH, Sengupta M, Fogg LF, Block JA. Effects of specialized footwear on joint loads in osteoarthritis of the knee. Arthritis Rheum. 2008 Sep 15;59(9):1214-20. doi: 10.1002/art.24017. PMID 18759313
- [Background] Shakoor N, Block JA. Walking barefoot decreases loading on the lower extremity joints in knee osteoarthritis. Arthritis Rheum. 2006 Sep;54(9):2923-7. doi: 10.1002/art.22123. PMID 16947448
- [Background] Shakoor N, Lidtke RH, Wimmer MA, Mikolaitis RA, Foucher KC, Thorp LE, Fogg LF, Block JA. Improvement in knee loading after use of specialized footwear for knee osteoarthritis: results of a six-month pilot investigation. Arthritis Rheum. 2013 May;65(5):1282-9. doi: 10.1002/art.37896. PMID 23575871